CLINICAL TRIAL: NCT01998815
Title: Role and Mechanisms of Obesity Surgery - Physical Activity and Other Predictors of Hospital Stay, Recovery and Complications After Obesity Surgery
Brief Title: Role and Mechanisms of Obesity Surgery
Acronym: RAMOSPHYSSURG
Status: Suspended | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: Dnr 310-13
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Obesity; Bariatric Surgery; Physical Activity; Post-operative Complications; Quality of Life
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obese patients: Laparoscopic Roux-en-Y gastric bypass
  Interventions: Procedure: Laparoscopic Roux-en-Y gastric bypass surgery

INTERVENTIONS:
Procedure: Laparoscopic Roux-en-Y gastric bypass surgery

SUMMARY:
The purpose of this study is to examine how physical activity and lifestyle factors influence postoperative recovery and postoperative complications after bariatric surgery.

The hypothesis is that physically active people, with a healthy alcohol consumption and non smokers have shorter lengths of hospital stay, shorter sick-leave, fewer re-hospitalizations and fewer re-operations, fewer complications as well as a faster recovery after a surgical procedure.

The investigators also hypothesize that possible risk factors for non-surgical postoperative complications e g abdominal discomfort are also life-style related factors such as smoking, high alcohol consumption, low level of physical activity, as well as other risk factors such as prior frequent abdominal pains (e g irritable bowel syndrome symptoms), high levels of anxiety and/or depression, difficulties with coping with the changed food intake regimen after obesity surgery, and generally high sensitivity for painful-sensations and nausea.

First aim of this study is to investigate how life style factors prior to obesity surgery are related to hospital stay, sick-leave, immediate postoperative complication rates and the rate of resumption of QoL and normal physical function.

The second aim of the study is to identify risk factors for the development of chronic abdominal discomfort and dumping symptoms after obesity surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 y of age
* BMI >35

Exclusion Criteria:

* non-knowledgeable in Swedish language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All obese patients undergoing laparoscopic Roux-en-Y gastric bypass surgery at Sahlgrenska University Hospital in Gothenburg and Kärnssjukhuset in Skövde, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative recovery and complications | 30 days
  Length of hospital stay, post-operative sick-leave, rate of post-operative complications; bleeding, anastomotic leakage, re-admission, re-operation, thromboembolic complications (deep-venous thrombosis, pulmonary embolism).

SECONDARY OUTCOMES:
Post-operative well-being and late complications | 24 months
  Post-operative well-being and late complications such as persistent gastrointestinal adverse symptoms abdominal discomfort, pain (measured using gastrointestinal symptom rating scale ;GSRS), dumping syndrome (measured by dumping syndrome rating scale), quality of life (SF-36 and EQ5d), physical activity level (Saltin Grimby), depression and anxiety rating (Hospital Depression and Anxiety rating scale), pain anxiety (Pain Catastrophizing scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Sahglrenska University Hospital, Gothenburg, Sweden